CLINICAL TRIAL: NCT06198933
Title: The Assessment of Hemolysis and Renal Functions During and After Catheter Ablation for Atrial Fibrillation Using Pulsed-field Energy
Brief Title: Renal Function and Hemolysis After Pulsed-field Ablation for Atrial Fibrillation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Sponsor
Other Study IDs: PFA RENAL HEMOLYSIS
Record Dates: First submitted 2023-12-28; First posted 2024-01-10 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2023-12

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; pulsed-fied ablation; hemolysis; renal function
MeSH Terms: conditions — Atrial Fibrillation; Hemolysis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples for the assessment of hemolysis and renal functions
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Pulsed-field ablation group: Patient with atrial fibrillation will undergo catheter ablation using pulsed-field energy
  Interventions: Device: Pulsed-field ablation

INTERVENTIONS:
Device: Pulsed-field ablation — Patients will atrial fibrillation will undergo catheter ablation using pulsed-field energy

SUMMARY:
The aim of the project is to assess hemolysis and renal function after catheter ablation for atrial fibrillation using pulsed-field energy. Hemolysis will be determined using the concentration of red blood cell microparticles at the end of the ablation (when all ablation were done, before sheath removal). Hemoglobinuria will be assessed one day after the procedure. Renal functions will be assessed one and three day after the procedure using standard parameters (creatinine, urea). The goal is to assess the acute worsening fo renal functions after pulsed-field ablation in relation to the number of PF applications, and to the degree of immediate post-procedural hemolysis.

DETAILED DESCRIPTION:
Methods The project will include patients with paroxysmal and persistent AF who, according to standard recommended procedures, are indicated for catheter ablation using pulsed-field energy and will sign informed consent. Patients with spontaneously present hemolysis (hematologic disorders) and patients in a dialysis program will be excluded. The catheterization procedure will be performed routinely as currently practiced at our institution. Specifically, pulmonary vein isolation will be conducted in all patients, and for patients with non-paroxysmal AF, additional additive ablation lesions will also be performed (most commonly ablation of the posterior wall of the left atrium and mitral isthmus, possibly the cavotricuspid isthmus). The ablation will always be performed under moderate sedation or general anesthesia with the participation of an anesthesiologist, as per our institution's practice. A total of 100 patients are planned to be enrolled. Prior to the procedure, patients will receive at least 4 weeks of anticoagulant treatment with NOACs, as recommended, and this treatment will be discontinued on the day of the procedure (i.e., the last tablet will be taken the day before the procedure). NOACs will be reintroduced into their medication regimen the day after ablation. All patients will undergo outpatient baseline blood tests, including renal function (creatinine, urea), as currently standard and required (up to 2 weeks before the procedure). Post-procedure, patients will be adequately hydrated; in addition to the recommended active oral intake post-procedure, all patients will receive an extra 1000 ml of saline solution during the afternoon following the procedure (unless there is a risk of overhydration, for instance, in the case of severe dysfunction).

Blood sampling Blood samples will be collected at two different times. Firstly, at the end of the procedure, 12 ml of blood will be drawn into tubes for hemolysis examination (anticoagulated blood with EDTA and Li-heparin). The degree of hemolysis will be assessed by examining red blood cell fragments (RBC microparticles) using flow cytometry. This examination is highly sensitive and capable of detecting even minimal amounts of damaged erythrocytes. The second blood sample will be collected the morning after the procedure, following the standard protocol, and will also include renal parameters (creatinine, urea) as routinely done. Additionally, on this day, a urine test for the presence of hemoglobinuria will be conducted. Both initial blood samples will be collected and analyzed during the hospitalization. A third sample for a follow-up assessment of kidney function will be required 2-3 days after the procedure. The patient will be asked to come either to our hospital for blood collection or to have it done at a laboratory near their residence. Results of this examination, if conducted outside the hospital, will be obtained from the patient over the phone. If kidney function in this sample is slightly reduced, the patient will be instructed for further monitoring or outpatient examination. In case of significantly elevated values, appropriate action will be advised promptly.

Three months post-procedure, an outpatient check-up will be conducted. Before this evaluation, the effectiveness of the ablation will be assessed using a 24-hour ECG Holter monitor, which is our current standard procedure. Additionally, kidney function will be rechecked. The purpose is to compare the number of applications of pulsed-field energy with the degree of hemolysis observed immediately after the procedure, along with kidney function shortly after. Hemolysis, the damage or breakdown of red blood cells, will be determined using a highly sensitive method and is practically certain to be present at the end of the procedure. However, whether hemolysis might lead to hemoglobinuria the following day in some cases has not been investigated, nor has the potential for temporary worsening of kidney function in certain patients. If this were the case, selecting at-risk patients (those with higher creatinine levels before the procedure) and implementing simple measures (sufficient fluid intake) could effectively prevent this complication. Our primary hypothesis is that while ablation using pulsed-field is associated with intravascular hemolysis, leading to the damage of some red blood cells, this process in only a minimal number of patients will result in hemoglobinuria, and it will not have any significant consequences on kidney function post-procedure.

ELIGIBILITY:
Inclusion Criteria:

* symptomatic paroxysmal or non-paroxysmal atrial fibrillation

Exclusion Criteria:

* known hematologic disorders
* disorders associated with increased hemolysis
* known significant hepatic disease
* patient in permanent hemodialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient will symptomatic paroxysmal or non-paroxysmal atrial fibrillation indicated for catheter ablation according to the standard criteria will be enrolled.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Red blood cell microparticles | day of the procedure - at the end of the procedure
  The concentration of red blood cell microparticles in the plasma assessed using flow cytometry
Hemoglobinuria | One day after the procedure
  The concentration of hemoglobin in urine
Creatinine three days | 3 days after the procedure
  The concentration of creatinine three days after ablation

SECONDARY OUTCOMES:
Lactate dehydrogenase | the day of the procedure - at the end of the procedure
  The concentration of lactate dehydrogenase at the end of ablation
Haptoglobin | the day of the procedure - at the end of the procedure
  The concentration of haptoglobin at the end of ablation
Creatinine one day | one day after the procedure
  The concentration of creatinine one day after ablation

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiocenter, 3rd Medical School, Charles University and University Hospital Kralovske Vinohrady, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No
Data will be shared 6 months after publication on request.

REFERENCES:
- [Background] Zoni-Berisso M, Filippi A, Landolina M, Brignoli O, D'Ambrosio G, Maglia G, Grimaldi M, Ermini G. Frequency, patient characteristics, treatment strategies, and resource usage of atrial fibrillation (from the Italian Survey of Atrial Fibrillation Management [ISAF] study). Am J Cardiol. 2013 Mar 1;111(5):705-11. doi: 10.1016/j.amjcard.2012.11.026. Epub 2012 Dec 28. PMID 23273528
- [Background] Wolf PA, Benjamin EJ, Belanger AJ, Kannel WB, Levy D, D'Agostino RB. Secular trends in the prevalence of atrial fibrillation: The Framingham Study. Am Heart J. 1996 Apr;131(4):790-5. doi: 10.1016/s0002-8703(96)90288-4. No abstract available. PMID 8721656
- [Background] Reddy VY, Dukkipati SR, Neuzil P, Anic A, Petru J, Funasako M, Cochet H, Minami K, Breskovic T, Sikiric I, Sediva L, Chovanec M, Koruth J, Jais P. Pulsed Field Ablation of Paroxysmal Atrial Fibrillation: 1-Year Outcomes of IMPULSE, PEFCAT, and PEFCAT II. JACC Clin Electrophysiol. 2021 May;7(5):614-627. doi: 10.1016/j.jacep.2021.02.014. Epub 2021 Apr 28. PMID 33933412
- [Background] Ekanem E, Reddy VY, Schmidt B, Reichlin T, Neven K, Metzner A, Hansen J, Blaauw Y, Maury P, Arentz T, Sommer P, Anic A, Anselme F, Boveda S, Deneke T, Willems S, van der Voort P, Tilz R, Funasako M, Scherr D, Wakili R, Steven D, Kautzner J, Vijgen J, Jais P, Petru J, Chun J, Roten L, Futing A, Rillig A, Mulder BA, Johannessen A, Rollin A, Lehrmann H, Sohns C, Jurisic Z, Savoure A, Combes S, Nentwich K, Gunawardene M, Ouss A, Kirstein B, Manninger M, Bohnen JE, Sultan A, Peichl P, Koopman P, Derval N, Turagam MK, Neuzil P; MANIFEST-PF Cooperative. Multi-national survey on the methods, efficacy, and safety on the post-approval clinical use of pulsed field ablation (MANIFEST-PF). Europace. 2022 Sep 1;24(8):1256-1266. doi: 10.1093/europace/euac050. PMID 35647644